CLINICAL TRIAL: NCT01310452
Title: A Multi-centre, Open-labeled, Randomized, Parallel Study on Liver Fat Content and Visceral Fat Mass in Overweight and Obese Type 2 Diabetes Patients After 26 Weeks Treatment With Insulin Detemir Once Daily Versus Insulin NPH Once Daily
Brief Title: Study on Liver Fat Content and Visceral Fat Mass in Overweight and Obese Type 2 Diabetes Patients After Treatment With Basal Insulin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Gao Xin/Professor, Department of Endocrinology and Metabolism, Zhongshan Hospital, Fudan University, Shanghai 200032 China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: prof gao xin
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes, basal insulin, metformin, liver fat, visceral fat
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Fatty Liver | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neutral protamine insulin, metformin (Active Comparator): NPH insulin once daily plus oral metformin twice or thrice daily during 26 weeks
  Interventions: Drug: insulin detemir
- insulin detemir, metformin (Experimental): Insulin detemir once daily plus oral metformin twice or thrice daily during 26 weeks
  Interventions: Drug: neutral protamine insulin

INTERVENTIONS:
Drug: insulin detemir — insulin detemir once daily with metformin
  Arms: neutral protamine insulin, metformin
Drug: neutral protamine insulin — neutral protamine insulin once daily with metformin
  Arms: insulin detemir, metformin

SUMMARY:
Primary objective:

To compare the change in liver fat content and visceral fat mass (cm2) assessed by MRS (Magnetic Resonance Spectroscopy) and MRI (Magnetic Resonance Image), after 26 weeks of treatment with insulin detemir once daily or insulin NPH once daily both with metformin in overweight and obese type 2 diabetic subjects.

Secondary objectives:

To compare the two treatments with respect to:

1. Efficacy:

   * MRI: abdominal subcutaneous fat mass(cm2), Calculated Visceral/Subcutaneous Adipose Tissue Ratio.
   * Change in HbA1c from baseline at 12 and 26 weeks of treatment.
   * Change in Fasting plasma glucose from baseline at 12 and 26 weeks of treatment.
   * Weight
   * Waist and hip circumference
2. Safety:

   * Incidence of hypoglycaemia in the 26 weeks of treatment with insulin detemir versus NPH
   * Lipid profile at the start and after 26 weeks of treatment
   * Incidence of Adverse events during the trial
   * Safety profile as measured by laboratory safety parameters (haematology, biochemistry) and physical examination/vital signs before and at the end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Female or male, 18 years≤age≤70years
* Subjects with insulin naïve type 2 diabetes who have been treated with metformin（>1g/d）alone for at least 3 months prior to screening
* 11%≥HbA1c≥7.5% based on analysis from a central laboratory
* 24kg/m2≤BMI≤40kg/m2
* Weight fluctuation<2kg in one month prior to screening
* Able and willing to perform self-monitoring of blood glucose.
* Willing to accept basal insulin therapy
* Able to self-inject all required doses of insulin

Exclusion Criteria:

* Treatment with any OADs (Oral Antidiabetic Drugs) in the last 6 months, except metformin (subjects currently treated with metformin within the interval of 1000-2000 mg daily may be included in the trial. The dose should have remained unchanged for a period of one month prior to randomisation and should be expected to remain unchanged throughout the trial period).
* Use of approved weight lowering pharmacotherapy (e.g. orlistat, sibutramine, rimonabant) or obesity induced by drug treatment (e.g. corticosteroids, NSAIDs, tricyclic anti-depressants, atypical anti-psychotics).
* Participation in a clinical study of weight control within the last 3 months prior to screening.
* Previous or planned surgical treatment of obesity.
* Any disease or condition (such as renal, hepatic or cardiac) according to the judgment of the Investigator makes the subject unsuitable for participation in the trial.
* Anticipated change in concomitant medication known to interfere with glucose metabolism, such as systemic steroids, non-selective beta-blockers or mono amine oxidase (MAO) inhibitors.
* Anticipated change in concomitant medication known to interfere with lipid metabolism, such as lipid-lowering drugs.
* Proliferative retinopathy or maculopathy that has required acute treatment within the last six months.
* Uncontrolled hypertension (treated or untreated) as judged by the Investigator
* Known or suspected allergy to trial product(s) or related products.
* Previous participation in this trial. Participation is defined as screened.
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures. Adequate contraceptive measures are sterilisation, intrauterine device (IUD), oral contraceptives or consistent use of barrier methods.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Any condition that the Investigator feels would interfere with trial participation or evaluation of results.
* Receipt of any investigational drug (NPH or insulin detemir) within 1 month prior to this trial.
* Cardiac disease defined according to NYHA class III or IV, unstable angina pectoris and/or myocardial infarction within the last 6 months previous to the selection.
* History of hypoglycaemic unawareness.
* With mental implant (such as cardiac pacemaker, insulin pump) in vivo.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
The change in liver fat content and visceral fat mass | After 26 weeks of treatment
  To compare the change in liver fat content and visceral fat mass (cm2), assessed by MRS and MRI, after 26 weeks of treatment with insulin detemir or insulin NPH (both with metformin) in overweight and obese type 2 diabetic subjects

SECONDARY OUTCOMES:
MRI | after 26 weeks of treatment
  Abdominal subcutaneous fat mass(cm2), Calculated Visceral/Subcutaneous Adipose Tissue Ratio.
Change in HbA1c | from baseline to 12 and 26 weeks of treatment respectively
  Change in HbA1c from baseline at 12 and 26 weeks of treatment respectively
Change in Fasting plasma glucose | From baseline to 12 and 26 weeks
  Change in Fasting plasma glucose (FPG) from baseline at 12 and 26 weeks of treatment respectively
Weight at every visit | At every visit
  Weight at every visit
Waist and hip circumference at every visit | At every visit
  Waist and hip circumference at every visit
Hypoglycaemia | during the 26-week treatment
  Incidence of hypoglycaemia in the 26 weeks of treatment with insulin detemir versus NPH
Lipid profile | At the start and after 26 weeks of treatment
  Lipid profile at the start and after 26 weeks of treatment
Adverse events | During the trial
  Incidence of Adverse events during the trial
Safety profile | During the treatment
  Safety profile as measured by laboratory safety parameters (haematology, biochemistry) and physical examination/vital signs before and at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Shan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Mokdad AH, Ford ES, Bowman BA, Nelson DE, Engelgau MM, Vinicor F, Marks JS. Diabetes trends in the U.S.: 1990-1998. Diabetes Care. 2000 Sep;23(9):1278-83. doi: 10.2337/diacare.23.9.1278. PMID 10977060
- [Background] Lean ME, Powrie JK, Anderson AS, Garthwaite PH. Obesity, weight loss and prognosis in type 2 diabetes. Diabet Med. 1990 Mar-Apr;7(3):228-33. doi: 10.1111/j.1464-5491.1990.tb01375.x. PMID 2139394
- [Background] Hollander P, Raslova K, Skjoth TV, Rastam J, Liutkus JF. Efficacy and safety of insulin detemir once daily in combination with sitagliptin and metformin: the TRANSITION randomized controlled trial. Diabetes Obes Metab. 2011 Mar;13(3):268-75. doi: 10.1111/j.1463-1326.2010.01351.x. PMID 21205123
- [Background] Whittingham JL, Havelund S, Jonassen I. Crystal structure of a prolonged-acting insulin with albumin-binding properties. Biochemistry. 1997 Mar 11;36(10):2826-31. doi: 10.1021/bi9625105. PMID 9062110
- [Background] Philis-Tsimikas A, Charpentier G, Clauson P, Ravn GM, Roberts VL, Thorsteinsson B. Comparison of once-daily insulin detemir with NPH insulin added to a regimen of oral antidiabetic drugs in poorly controlled type 2 diabetes. Clin Ther. 2006 Oct;28(10):1569-81. doi: 10.1016/j.clinthera.2006.10.020. PMID 17157113
- [Background] Mandosi E, Fallarino M, Rossetti M, Gatti A, Morano S. Waist circumference reduction after insulin detemir therapy in type 2 diabetes patients previously treated with NPH. Diabetes Res Clin Pract. 2009 May;84(2):e18-20. doi: 10.1016/j.diabres.2009.02.006. Epub 2009 Mar 17. PMID 19297054
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419